CLINICAL TRIAL: NCT07393009
Title: Observation of Clinical Routine Care for Patients Implanted With BIOTRONIK Devices Used for Conduction System Pacing (CSP)
Brief Title: Studying Routine Patient Care With BIOTRONIK Devices That Allow a More Natural Heart Stimulation
Acronym: BIO|STREAM-CSP
Status: Not yet recruiting | Type: Observational
Sponsor: Biotronik SE & Co. KG (Industry)
Responsible Party: Sponsor
Other Study IDs: BA118
Record Dates: First submitted 2026-01-09; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2025-12

CONDITIONS: Cardiac Pacing; Cardiac Pacemaker; Implantable Cardioverter Defibrillator; Cardiac Resynchronization Therapy Devices; Bradycardia; Tachycardia; Heart Failure
Keywords: Conduction system pacing (CSP); Left bundle branch area pacing (LBBAP)
MeSH Terms: conditions — Bradycardia; Tachycardia; Heart Failure

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 4 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Implantation of the Solia CSP S pacing lead for LBBAP — Observation of clinical routine care for patients implanted with BIOTRONIK devices used for conduction system pacing (CSP)

SUMMARY:
The registry is designed to assess outcome, performance and residual safety aspects of BIOTRONIK products which are used in the context of CSP based on long-term data from an unselected, real-life clinical set-up.

ELIGIBILITY:
Inclusion Criteria:

* Guideline indication for pacemaker or cardiac resynchronization therapy with or without defibrillation function (CRT-P/-D)
* Patient is intended for a de novo implantation and LBBAP therapy with an investigational generator and an investigational lead OR has just been implanted with an investigational generator and an investigational lead positioned permanently deep within the intraventricular septum and has not yet been discharged from the hospital OR transitions from the BIO|MASTER.CSP study
* Ability to understand the nature of the study
* Ability and willingness to perform all follow-up visits
* Ability and willingness to use the CardioMessenger and acceptance of the BIOTRONIK Home Monitoring concept

Exclusion Criteria:

* Planned dation from intended use
* Planned for cardiac surgical procedures, heart transplantation or interventional measures other than the study procedure within one year after enrollment
* Life-expectancy less than 12 months
* Pregnant or breast feeding
* Age less than 18 years
* Participation in an interventional clinical investigation, except for submodules within this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The patient population consists exclusively of patients with an indication for pacemaker or cardiac resynchronization therapy according to the current clinical practice.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2033-02-01 (Estimated); Study Completion 2033-02-01 (Estimated)

PRIMARY OUTCOMES:
SADE-d free rate related to any investigatonal device | throughout study duration, average of 4 years; annual evaluations
  Rate of serious adverse device effects possible, probable or causal related to any investigational device.
Rate of successful acute implantation in LBBAP using investigational devices in LBBAP | Day 1
  All implantations, in which the investigator decides to leave the Solia CSP S pacing lead permanently deep within the intraventricular septum are counted as acute success.
Capture type at implantation | Day 1
  The investigator confirms the type of pacing capture for any implantation in which the pacing lead is permanently positioned deep within the interventricular septum. Success rates for LBBAP and CSP are determined based on ECG parameters.
Long-term maintenance of LBBAP | throughout study duration, average of 4 years; annual evaluations
  The investigator is asked to assess the effectiveness of LBBAP during follow-up based on the interpretation of a 12-lead ECG recording.
Electrical parameters - pacing threshold | throughout study duration, average of 4 years; annual evaluations
  The investigators will be asked to record the pacing thresholds (Volts) of the LBBAP leads at a pulse width of 0.4 ms.
Electrical parameters - sensing amplitude | throughout study duration, average of 4 years; annual evaluations
  The investigators will be asked to record the sensing amplitude (Millivolts) of the LBBAP leads.
Electrical parameters - pacing impedance | throughout study duration, average of 4 years; annual evaluations
  The investigators will be asked to record the lead pacing impedance (Ohms) of the LBBAP leads.